CLINICAL TRIAL: NCT00455793
Title: Subclinical Atherosclerosis in HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2006-P-000238
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Coronary Atherosclerosis
Keywords: HIV; atherosclerosis
MeSH Terms: conditions — HIV Infections; Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: HIV
- 2: Non-HIV infected controls

SUMMARY:
We will obtain data using multi-slice CT technology to detect subclinical coronary disease in the HIV population. Determination of subclinical cardiovascular disease using noninvasive technology and elucidation of the associated risk factors will help to guide targeted therapy to prevent cardiovascular events in this patient population.

We will investigate the prevalence of coronary plaque lesions and coronary artery calcifications in men and women with HIV disease as determined by 64-row multidetector computed tomography (MDCT) and MDCT coronary angiography in comparison to age-matched control subjects without HIV infection. We hypothesize that evidence of coronary artery calcification and coronary plaque lesions as seen by MDCT will be present in individuals with HIV more than non-HIV control subjects of the same age. We also hypothesize the degree of atherosclerosis will be increased in HIV patients compared to control subjects.

We will evaluate the metabolic and inflammatory factors associated with coronary artery disease in HIV-infected individuals. We hypothesize that traditional cardiac risk factors as well as metabolic and inflammatory changes associated with HIV and its treatment such as dyslipidemia, increased secretion of inflammatory markers, decreased adiponectin, increased insulin resistance and increased visceral fat may be associated with coronary artery disease in HIV-infected individuals.

ELIGIBILITY:
Inclusion criteria for HIV infected subjects arm:

1. Men and women age 18-60
2. BMI 20-35
3. Previously documented HIV disease for 5 years or longer either on stable highly active anti-retroviral therapy (HAART) or not on HAART.
4. No changes in antiretroviral regimen within the prior 3 months.

Inclusion criteria for non-HIV infected control subjects arm:

1. Healthy men and women age 18-60
2. BMI 20-35

Exclusion criteria for both arms:

1. Previously diagnosed coronary artery disease, cerebrovascular disease, or peripheral vascular disease.
2. Use of glucocorticoids, growth hormone, testosterone, or other anabolic agents within past 6 months
3. Renal disease or creatinine >1.5 mg/dL
4. Anti-inflammatory medications
5. Opportunistic infection within past 6 months in HIV infected individuals and current acute infectious illness in both HIV-infected subjects and normal controls.
6. Nitrates or others medications that can alter endothelial function
7. Contraindication to beta-blocker use
8. Body weight greater than 300 lbs due to DEXA scanner table limitations
9. Patients with previous allergic reactions to iodine-containing contrast media or to iodine will be excluded from participation
10. Active illicit drug use
11. Pregnancy or breastfeeding
12. Estrogen or progestin use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV infected men and women and non-HIV infected control men and women
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2006-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Coronary Plaque | Baseline

SECONDARY OUTCOMES:
Inflammatory indices, glucose homeostasis, body composition | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sim JH, Sherman JB, Stanley TL, Corey KE, Fitch KV, Looby SE, Robinson JA, Lu MT, Burdo TH, Lo J. Pro-Inflammatory Interleukin-18 is Associated with Hepatic Steatosis and Elevated Liver Enzymes in People with HIV Monoinfection. AIDS Res Hum Retroviruses. 2021 May;37(5):385-390. doi: 10.1089/AID.2020.0177. Epub 2021 Jan 25. PMID 33323025
- [Derived] Cheru LT, Saylor CF, Fitch KV, Looby SE, Lu M, Hoffmann U, Stanley TL, Lo J. Low vitamin D is associated with coronary atherosclerosis in women with HIV. Antivir Ther. 2019;24(7):505-512. doi: 10.3851/IMP3336. PMID 31742564
- [Derived] Fourman LT, Saylor CF, Cheru L, Fitch K, Looby S, Keller K, Robinson JA, Hoffmann U, Lu MT, Burdo T, Lo J. Anti-Inflammatory Interleukin 10 Inversely Relates to Coronary Atherosclerosis in Persons With Human Immunodeficiency Virus. J Infect Dis. 2020 Feb 3;221(4):510-515. doi: 10.1093/infdis/jiz254. PMID 31077265
- [Derived] Weiss JJ, Sanchez L, Hubbard J, Lo J, Grinspoon SK, Fitch KV. Diet Quality Is Low and Differs by Sex in People with HIV. J Nutr. 2019 Jan 1;149(1):78-87. doi: 10.1093/jn/nxy241. PMID 30624677
- [Derived] Cheru LT, Park EA, Saylor CF, Burdo TH, Fitch KV, Looby S, Weiner J, Robinson JA, Hubbard J, Torriani M, Lo J. I-FABP Is Higher in People With Chronic HIV Than Elite Controllers, Related to Sugar and Fatty Acid Intake and Inversely Related to Body Fat in People With HIV. Open Forum Infect Dis. 2018 Nov 5;5(11):ofy288. doi: 10.1093/ofid/ofy288. eCollection 2018 Nov. PMID 30515430
- [Derived] Srinivasa S, Fitch KV, Torriani M, Zanni MV, Defilippi C, Christenson R, Maehler P, Looby SE, Lo J, Grinspoon SK. Relationship of visceral and subcutaneous adipose depots to markers of arterial injury and inflammation among individuals with HIV. AIDS. 2019 Feb 1;33(2):229-236. doi: 10.1097/QAD.0000000000002060. PMID 30325779
- [Derived] Zanni MV, Stone LA, Toribio M, Rimmelin DE, Robinson J, Burdo TH, Williams K, Fitch KV, Lo J, Grinspoon SK. Proprotein Convertase Subtilisin/Kexin 9 Levels in Relation to Systemic Immune Activation and Subclinical Coronary Plaque in HIV. Open Forum Infect Dis. 2017 Oct 14;4(4):ofx227. doi: 10.1093/ofid/ofx227. eCollection 2017 Fall. PMID 29226174
- [Derived] Srinivasa S, Lu MT, Fitch KV, Hallett TR, O'Malley TK, Stone LA, Martin A, Coromilas AJ, Burdo TH, Triant VA, Lo J, Looby SE, Neilan TG, Zanni MV. Epicardial adipose tissue volume and cardiovascular risk indices among asymptomatic women with and without HIV. Antivir Ther. 2018;23(1):1-9. doi: 10.3851/IMP3193. PMID 28930079
- [Derived] Fitch KV, DeFilippi C, Christenson R, Srinivasa S, Lee H, Lo J, Lu MT, Wong K, Petrow E, Sanchez L, Looby SE, Hoffmann U, Zanni M, Grinspoon SK. Subclinical myocyte injury, fibrosis and strain in relationship to coronary plaque in asymptomatic HIV-infected individuals. AIDS. 2016 Sep 10;30(14):2205-14. doi: 10.1097/QAD.0000000000001186. PMID 27314177
- [Derived] Looby SE, Fitch KV, Srinivasa S, Lo J, Rafferty D, Martin A, Currier JC, Grinspoon S, Zanni MV. Reduced ovarian reserve relates to monocyte activation and subclinical coronary atherosclerotic plaque in women with HIV. AIDS. 2016 Jan 28;30(3):383-93. doi: 10.1097/QAD.0000000000000902. PMID 26696388
- [Derived] Zanni MV, Kelesidis T, Fitzgerald ML, Lo J, Abbara S, Wai B, Marmarelis E, Hernandez NJ, Yang OO, Currier JS, Grinspoon SK. HDL redox activity is increased in HIV-infected men in association with macrophage activation and non-calcified coronary atherosclerotic plaque. Antivir Ther. 2014;19(8):805-811. doi: 10.3851/IMP2756. Epub 2014 Feb 17. PMID 24535655
- [Derived] Fitch KV, Srinivasa S, Abbara S, Burdo TH, Williams KC, Eneh P, Lo J, Grinspoon SK. Noncalcified coronary atherosclerotic plaque and immune activation in HIV-infected women. J Infect Dis. 2013 Dec 1;208(11):1737-46. doi: 10.1093/infdis/jit508. Epub 2013 Sep 16. PMID 24041790
- [Derived] Hwang JJ, Wei J, Abbara S, Grinspoon SK, Lo J. Receptor activator of nuclear factor-kappaB ligand (RANKL) and its relationship to coronary atherosclerosis in HIV patients. J Acquir Immune Defic Syndr. 2012 Nov 1;61(3):359-63. doi: 10.1097/QAI.0b013e31826a6c16. PMID 22842843
- [Derived] Burdo TH, Lo J, Abbara S, Wei J, DeLelys ME, Preffer F, Rosenberg ES, Williams KC, Grinspoon S. Soluble CD163, a novel marker of activated macrophages, is elevated and associated with noncalcified coronary plaque in HIV-infected patients. J Infect Dis. 2011 Oct 15;204(8):1227-36. doi: 10.1093/infdis/jir520. PMID 21917896
- [Derived] Lo J, Abbara S, Rocha-Filho JA, Shturman L, Wei J, Grinspoon SK. Increased epicardial adipose tissue volume in HIV-infected men and relationships to body composition and metabolic parameters. AIDS. 2010 Aug 24;24(13):2127-30. doi: 10.1097/QAD.0b013e32833c055a. PMID 20588167